CLINICAL TRIAL: NCT03368989
Title: The Effects of Radium-223 Dichloride Therapy on Radionuclide Bone Scan Lesions.
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Isis W Gayed, Professor, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-14-0113
Record Dates: First submitted 2017-11-13; First posted 2017-12-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Bony Metastases From Castrate Refractory Prostate Cancer
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- treatment with radium-223 Dichloride (Xofigo)
  Interventions: Drug: Radium-223 dichloride

INTERVENTIONS:
Drug: Radium-223 dichloride — Previously known as Alpharadin, Radium-223 dichloride is a calcium-mimetic, alpha emitting radiopharmaceutical, which introduces double-stranded DNA breaks in metastatic cancer cells.
  Other Names: Xofigo

SUMMARY:
To describe the changes seen on bone scan and correlate them with changes in relative chemical biomarkers, patient's functional status and level of pain.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients scheduled for treatment with Radium-223.

Exclusion Criteria:

* Patients not completing their treatment regimen for any reason

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males presenting with prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Change in number of osteoblastic bone lesions | Pretreatment (about 30 days before treatment) and post treatment (about 4 weeks after treatment)
  number of lesions specified before and after the treatment with a bone scan

SECONDARY OUTCOMES:
functional status as indicated by score on the Eastern Cooperative Oncology Group (ECOG) performance scale | Pretreatment (about 1 to 3 days before each treatment) for a total of 6 treatments
  The ECOG scale describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability (walking, working, etc.). The possible scores on the scale are 0 to 5, with 0 being the best outcome and 5 being the worst outcome, details of each score are listed below.
  Grade 0 = Fully active, able to carry on all pre-disease performance without restriction Grade 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work Grade 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours Grade 3 = Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours Grade 4 = Completely disabled; cannot carry on any selfcare; totally confined to bed or chair Grade 5 = Dead
pain level as assessed by numeric rating score | Pretreatment (about 1 to 3 days before each treatment) for a total of 6 treatments
  As assessed using numeric rating score from 1-10 with 10 being the highest level of pain
(PSA) prostate specific antigen level | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  normal level should be 4.0 ng/mL. value is measured after each dose
(ALP) alkaline phosphatase level | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  The normal value for alkaline phosphatase is 53 to 128 U/L.
Hemoglobin level | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  The normal level for males is 14 to 18 g/dl
Platelet level | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  A normal platelet count ranges from 150,000 to 450,000 platelets
Neutrophil count | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  The normal range for neutrophils is 2.5-7.5 x 10 9 /L
Creatinine level | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  Normal levels of creatinine in the blood are approximately 0.6 to 1.2 milligrams (mg) per deciliter (dL)
white blood cell count | pretreatment (about 1 to 7 days before each treatment) for a total of 6 treatments
  The typical white blood cell count varies from 4,000 to 10,000 cells per mm3.

CONTACTS AND LOCATIONS:
Overall Officials: Isis W Gayed, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No